CLINICAL TRIAL: NCT05041179
Title: Investigation on the Bioavailability of PRUVIN® and Its Effects on Physiologic-metabolic Biomarkers in Healthy Subjects
Brief Title: Bioavailability of PRUVIN® and Its Effects in Healthy Subjects (INDIGO)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Société des Produits Nestlé (SPN) (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Other
Other Study IDs: 18.01.CLI
Record Dates: First submitted 2021-09-02; First posted 2021-09-10 (Actual); Last update posted 2024-10-22 (Actual); Status verified 2024-10

CONDITIONS: Oxidative Stress
Keywords: Glutathione
MeSH Terms: interventions — isomaltulose

STUDY DESIGN:
Intervention Model Description: Double-blind, randomized, Placebo-controlled
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- 7.2 g of actives (3.6 g NAC and 3.6 g glycine) per day split in two doses (arm A) (Active Comparator): * First dose (1.8 g NAC and 1.8 g glycine) consumed in the morning
  * Second dose (1.8 g NAC and 1.8 g glycine) taken in the evening
  Interventions: Dietary Supplement: Pruvin R
- 4.8 g of actives (2.4 g NAC and 2.4 g glycine) per day split in two doses (arm B) (Active Comparator): * First dose (1.2 g NAC and 1.2 g glycine, +1.2 g placebo) consumed in the morning
  * Second dose (1.2 g NAC and 1.2 g glycine, +1.2 g placebo) taken in the evening
  Interventions: Dietary Supplement: Pruvin R
- 2.4 g of actives (1.2 g NAC and 1.2 g glycine) per day split in two doses (arm C) (Active Comparator): * First dose (0.6 g NAC and 0.6 g glycine, +2.4 g placebo) consumed in the morning
  * Second dose (0.6 g NAC and 0.6 g glycine, +2.4 g placebo) taken in the evening
  Interventions: Dietary Supplement: Pruvin R
- Placebo control (7.2 g isomaltulose)(arm D) (Placebo Comparator): * First dose (3.6 g isomaltulose) consumed in the morning
  * Second dose (3.6 g isomaltulose) taken in the evening
  Interventions: Other: Isomaltulose

INTERVENTIONS:
Dietary Supplement: Pruvin R — Combination of N-acetylcysteine an glycine
  Arms: 2.4 g of actives (1.2 g NAC and 1.2 g glycine) per day split in two doses (arm C); 4.8 g of actives (2.4 g NAC and 2.4 g glycine) per day split in two doses (arm B); 7.2 g of actives (3.6 g NAC and 3.6 g glycine) per day split in two doses (arm A)
Other: Isomaltulose — Placebo as comparator to intervention
  Arms: Placebo control (7.2 g isomaltulose)(arm D)

SUMMARY:
To evaluate the effect of different doses of PRUVIN® (N-acetylcysteine [NAC] and glycine) on reduced glutathione levels in healthy elderly subjects

DETAILED DESCRIPTION:
This is a single-center, double-blind, randomized, placebo-controlled 4-arm study-design, to assess the safety, tolerability and effect of PRUVIN® on reduced glutathione levels in healthy elderly (age 60-85 years) subjects.

In addition, baseline values of glutathione precursors, glutathione, and plasma markers of oxidative stress in a healthy young cohort (non-interventional) will be compared with those of the healthy elderly cohort (interventional).

ELIGIBILITY:
Non-interventional cohort:

Inclusion criteria:

1. 20-40 years, both inclusive
2. male and female
3. Considered generally healthy upon completion of medical history and screening safety assessments, as judged by the Investigator.
4. BMI >18.5 and <30.0 kg/m2
5. HbA1c <5.7 %
6. Informed consent as documented by signature

Exclusion criteria:

1. Receipt of any medicinal product or nutritional product in clinical development within 30 days before enrollment in this trial.
2. Any history or presence of clinically relevant comorbidity, as judged by the Investigator.
3. Signs of acute illness as judged by the Investigator.
4. Any serious systemic infectious disease during four weeks prior enrollment in this trial
5. Clinically significant abnormal screening laboratory tests, as judged by the Investigator.
6. AST and/or ALT > 2 times the upper limit of normal.
7. Elevated serum creatinine values above the upper limit of normal.
8. Systolic blood pressure < 90 mmHg or >139 mmHg and/or diastolic blood pressure < 50 mmHg or >89 mmHg (excluding white-coat hypertension; therefore, a repeat test showing results within range will be acceptable).
9. Heart rate at rest outside the range of 50-90 beats per minute.
10. Clinically significant abnormal standard 12-lead electrocardiogram (ECG) after 5 minutes resting in supine position at screening, as judged by the Investigator.
11. Significant history of alcoholism or drug abuse as judged by the Investigator consuming more than 24 grams alcohol/day (for males), 12 grams alcohol/day (for females) on average.
12. Smoking or use of nicotine substitute products.
13. Any medication (prescription and non-prescription drugs) within 14 days before screening.
14. Blood donation or blood loss of more than 500 mL within the last 3 months prior to screening.
15. Mental incapacity, unwillingness or language barriers precluding adequate understanding or co-operation.
16. If female, pregnant or breast-feeding.
17. Consumption of high protein supplements within 60 days of screening and during the study.
18. Consumption of any antioxidant, vitamins, and herbals (see chapter 12.2) supplements within 2 weeks prior to screening and during the study.

Interventional Cohort:

Inclusion Criteria:

1. 60-85 years, both inclusive
2. male and female
3. Sedentary, less than 1h of strenuous physical exercise per week
4. BMI of 25.0 to 35.0 kg/m2, both inclusive
5. HbA1c<6.5 %
6. Informed consent as documented by signature

Exclusion Criteria:

1. Known or suspected hypersensitivity to any component of the trial products.
2. Receipt of any medicinal product or nutritional product in clinical development within 30 days before randomisation in this trial.
3. History of multiple and/or severe allergies to drugs or foods or a history of severe anaphylactic reaction.
4. Any history or presence of clinically relevant comorbidity, as judged by the Investigator.
5. Signs of acute illness as judged by the Investigator.
6. Any serious systemic infectious disease during four weeks prior to first intake of the trial product, as judged by the Investigator.
7. Clinically significant abnormal screening laboratory tests, as judged by the Investigator.
8. AST and/or ALT > 2 times the upper limit of normal.
9. Elevated serum creatinine values above the upper limit of normal.
10. Systolic blood pressure < 90 mmHg or >139 mmHg and/or diastolic blood pressure < 50 mmHg or >89 mmHg (excluding white-coat hypertension; therefore, a repeat test showing results within range will be acceptable).
11. Heart rate at rest outside the range of 50-90 beats per minute.
12. Clinically significant abnormal standard 12-lead electrocardiogram (ECG) after 5 minutes resting in supine position at screening, as judged by the Investigator.
13. Significant history of alcoholism or drug abuse as judged by the Investigator consuming more than 24 grams alcohol/day (for males), 12 grams alcohol/day (for females) on average.
14. Smoking more than 5 cigarettes or the equivalent per day.
15. Inability or unwillingness to refrain from smoking and use of nicotine substitute products 3 days prior and during the intervention.

Ages: 20 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 128 (Actual)
Dates: Start 2019-04-01 (Actual); Primary Completion 2020-04-01 (Actual); Study Completion 2020-05-01 (Actual)

PRIMARY OUTCOMES:
Total reduced glutathione | 2 weeks
  Total reduced glutathione (GSH-T) in whole-blood normalized to hematocrit

SECONDARY OUTCOMES:
Free reduced glutathione | 2 weeks
  Free reduced glutathione (GSH-F), free reduced glutathione to oxidized glutathione disulfide ratio (GSH-F:GSSG)
Hematocrit | 2 weeks
  Whole-blood concentrations of glycine and cysteine normalized to hematocrit
Lipid oxidation | 2 weeks
  Lipid oxidation derived from indirect calorimetry

CONTACTS AND LOCATIONS:
Overall Officials: Ulrike Hövelmann, MD, Principal Investigator — Profil Institut für Stoffwechselforschung GmbH
Locations (1):
- Profil Institut für Stoffwechselforschung GmbH, Neuss, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Lizzo G, Migliavacca E, Lamers D, Frezal A, Corthesy J, Vinyes-Pares G, Bosco N, Karagounis LG, Hovelmann U, Heise T, von Eynatten M, Gut P. A Randomized Controlled Clinical Trial in Healthy Older Adults to Determine Efficacy of Glycine and N-Acetylcysteine Supplementation on Glutathione Redox Status and Oxidative Damage. Front Aging. 2022 Mar 7;3:852569. doi: 10.3389/fragi.2022.852569. eCollection 2022. PMID 35821844